CLINICAL TRIAL: NCT01743339
Title: A Randomized Controlled Trial of CBT for Insomnia in Patients With PTSD and Depression
Brief Title: Managing Sleep Symptoms and Modifying Mechanisms of Traumatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Wilfred Pigeon, PhD, Associate Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44033; R01NR013909 (NIH)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2016-08

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Sleep
Keywords: Randomized Controlled Trial; Cognitive Therapy; Stress Disorders, Post-Traumatic; Depression; Sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Control (brief check-in calls) and Cognitive Processing Therapy (12 individual weekly sessions)
  Interventions: Behavioral: Control
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy for Insomnia (4 individual therapy sessions over 5 weeks) and Cognitive Processing Therapy (12 individual weekly sessions)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy for Insomnia(4 individual therapy sessions over 5 weeks) will consist of a standard, structured, multi-component CBT intervention (sleep education, sleep hygiene, sleep restriction, stimulus control, cognitive therapy, and relapse prevention) Cognitive Processing Therapy will consist of a standard, structured 12-session protocol (PTSD education, exploring personal impact of trauma, experiencing emotions related to thoughts of trauma, cognitive therapy, and applying healthy thoughts and behaviors) delivered in individual weekly sessions
  Other Names: Cognitive-Behavioral Therapy for Insomnia; Cognitive Processing Therapy
  Arms: Cognitive Behavioral Therapy
Behavioral: Control — Cognitive Processing Therapy will consist of a standard, structured 12-session protocol (PTSD education, exploring personal impact of trauma, experiencing emotions related to thoughts of trauma, cognitive therapy, and applying healthy thoughts and behaviors) delivered in individual weekly sessions.
  Other Names: Cognitive Processing Therapy
  Arms: Control

SUMMARY:
The primary purpose of this study is to test whether and how cognitive-behavioral therapy for insomnia (CBTi), a well-supported and highly effective insomnia treatment, may directly improve Posttraumatic Stress Disorder (PTSD) and Major Depressive Disorder (MDD) symptoms. The study is designed as a randomized controlled trial (RCT) to test the effect of CBTi on symptoms of PTSD and co-morbid depression prior to an evidence-based PTSD intervention and to assess the role of neurobiological processes and sleep architecture in mediating treatment outcomes.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD), which occurs in at least 15-20% of individuals exposed to a traumatic event, is a chronic condition associated with the development of a multitude of negative physical and mental health consequences and the co-occurrence of Major Depressive Disorder (MDD). Sleep disturbances, and especially nightmares and insomnia, are quite common in patients with PTSD, but the standard treatments for PTSD do not directly focus on sleep problems. Perhaps as a result, sleep disturbances are one of the most common residual symptoms following both PTSD treatments and depression treatments. Importantly, insomnia, depression and PTSD are each characterized by similar biological dysregulation, including alterations in important aspects of sleep (rapid eye movement sleep and slow wave sleep) as well as processes linked to health and disease (stress system responses and inflammatory processes).

Directly treating sleep in the context of PTSD and MDD is feasible and can lead to robust improvements in sleep, though whether improving sleep can enhance PTSD and MDD outcomes remains to be established. This study will enroll and randomize 150 participants with PTSD, MDD and insomnia. Following baseline assessments (T1) participants will be randomized to receive cognitive-behavioral therapy for insomnia(CBTi), a well-supported and highly effective insomnia treatment, or to a monitor only control condition. Following this first intervention period all participants will receive cognitive processing therapy, a trauma focused therapy with known effects on PTSD and depression. The study will test whether and how CBTi may(1) achieve improvements in PTSD and MDD symptom severity and (2) lead to enhanced response to subsequent treatment with cognitive processing therapy.

Intervening with CBTi prior to a PTSD-specific treatment and measuring biomarkers longitudinally, will allow for the testing of specific effects of sleep improvement on PTSD, depressive symptoms, objective aspects sleep and stress and inflammatory markers, thereby advancing basic understanding of biobehavioral mechanisms in PTSD and depression. Importantly, the proposed approach utilizes a treatment sequence that may appeal to trauma survivors with post-traumatic event symptoms who may be resistant to or unprepared to fully engage in standard PTSD treatments. Confirmation of the study hypotheses could support immediate translation of the findings to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* must be English-speaking
* age 18-64 years old
* with exposure to trauma from interpersonal violence in the past year
* meet diagnostic criteria for full or subthreshold PTSD
* meet diagnostic criteria for MDD
* meet criteria for Insomnia Disorder

Exclusion Criteria:

* untreated sleep disorders other than insomnia or nightmares
* dementia or cognitive impairment
* history of schizophrenia or bipolar I disorder
* current suicidality
* health conditions with immunological components or taking immunosuppressive therapies
* active alcohol dependence
* medication use including antipsychotics, opiate analgesics, and sleep medications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2013-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
PTSD (intensity and frequency for each symptom, and remission) | 20 weeks
  The Clinician Administered PTSD Scale (CAPS)will be used as our primary PTSD outcome measure.

SECONDARY OUTCOMES:
Insomnia severity | 20 weeks
  The Insomnia Severity Index will measure insomnia severity.
Depression | 20 weeks
  The Hamilton Rating Scale for Depression-17 (HRSD-17)will be used as our primary measure of depressive symptoms. The MINI will be used to identify MDD remission status.

OTHER OUTCOMES:
Sleep | 7 weeks.
  The primary objective sleep outcomes will be rapid eye movement (REM) arousals and Slow Wave Activity.
Salivary Cortisol | 7 weeks
  Salivary cortisol will be measured in the Psychoneuroimmunology (PNI) Lab using a cortisol HS enzyme immunoassay kit.
Inflammatory cytokine levels (IL-6) | 7 weeks
  Inflammatory cytokine levels (IL-6) will be measured in the PNI Lab using Quantikine high sensitivity (HS) ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred R. Pigeon, Ph.D., Principal Investigator — University of Rochester; Kathi L. Heffner, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.

REFERENCES:
- [Derived] Pigeon WR, Heffner KL, Crean H, Gallegos AM, Walsh P, Seehuus M, Cerulli C. Responding to the need for sleep among survivors of interpersonal violence: A randomized controlled trial of a cognitive-behavioral insomnia intervention followed by PTSD treatment. Contemp Clin Trials. 2015 Nov;45(Pt B):252-260. doi: 10.1016/j.cct.2015.08.019. Epub 2015 Sep 4. PMID 26343743